CLINICAL TRIAL: NCT05469269
Title: Cleveland African American Prostate Cancer Project: Equivalence of Passive Navigation, Active Navigation, and Community-based Screening for Completion of Prostate Cancer Screening
Brief Title: Cleveland African American Prostate Cancer Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CASE7822
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analyst will be blinded to the study arm assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education and Passive Navigation (Experimental): This arm receives barber-led education and access to a resource website. Barbers will encourage clients to access the screening website. Other study materials will also be located within the shop. The resource website will be accessible via QR code that will encourage potential participants to complete a Prostate Cancer Knowledge and Risk Assessment questionnaire.
  Interventions: Behavioral: Passive Education
- Education and Active Navigation (Experimental): This arm includes all interventions of the first arm plus the addition of a community navigator. The community navigator will be onsite to assist in information delivery and navigation to resources and encourage the completion of the Screener through the QR code. The community navigator will help participants connect with a primary care provider to continue with all preventive healthcare recommendations.
  Interventions: Behavioral: Passive Education; Behavioral: Education by Community Navigator
- Education and Active Navigation with Community Based Outreach (Experimental): This arm adds the community navigator and a community outreach screening event. Case Comprehensive Cancer Center Community Outreach and Engagement will offer barber shops an onsite PSA screening event.
  Interventions: Behavioral: Passive Education; Behavioral: Education by Community Navigator; Behavioral: Education at Community Outreach Screening Event

INTERVENTIONS:
Behavioral: Passive Education — Education: QR codes will be posted at each barber's station within a barber shop, as well as on other study materials located within the shop. The QR code recruitment mechanism will encourage potential participants to complete a Prostate Cancer Knowledge and Risk Assessment questionnaire (ie. Screener) which acts as a screener for study eligibility. The screener can be completed by scanning the QR code with a cell phone while in the barbershop. Barbers will encourage their clients to complete the Screener.
Behavioral: Education by Community Navigator — A community navigator will be onsite to assist in information delivery, navigation to resources, and encourage the completion of the Screener through the QR code. Participants can opt to connect with the community navigator if they have questions, need assistance in scheduling a PSA screening, or if they have other resource needs. The community navigator will help participants connect with a primary care provider to continue with all preventive healthcare recommendations.
  Arms: Education and Active Navigation; Education and Active Navigation with Community Based Outreach
Behavioral: Education at Community Outreach Screening Event — The Community Navigator will set up PSA screening events at specific barber shops for participants who wish to move forward with screenings.
  Arms: Education and Active Navigation with Community Based Outreach

SUMMARY:
The purpose of this research is to test intervention strategies that encourage and support Black or African American men who are 40 and older to complete prostate cancer screening, and specifically to complete a prostate-specific antigen (PSA) test.

DETAILED DESCRIPTION:
This intervention is designed to evaluate the effectiveness of three different approaches to increasing PSA screening in African American men, starting at age 40. The approaches are 1) education and passive navigation, 2) education and active navigation, and 3) education and active navigation with community based outreach. Completion of a PSA blood test is the primary outcome of this study, which will be evaluated four months following the recruitment phase at each shop. At the 4 month follow-up, participants will be asked about PSA completion; participants who completed PSA screening will be asked to provide outcomes from their PSA screening (ie. PSA results and provider recommended next steps), as well as their feelings regarding their screening experience, trust in the screening process, and knowledge about prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years old
* Self-identify as Black or African American
* Have a prostate gland (includes biological males, transwomen)
* PSA-naïve or has not received a PSA test in the past 12 months
* Has not had a previous prostate cancer diagnosis
* English speaking
* Ability to consent to study

Exclusion Criteria:

* Individuals who have had a prostatectomy

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
PSA Screening Test | At 4 months
  The number of participants who had a PSA screening test completed.

SECONDARY OUTCOMES:
PSA Screening Test | At 14 months
  The number of participants who had a PSA screening test completed.
Primary Care Physician Visit | At 4 months
  The number of participants that followed up with a primary care physician for a visit or to establish long-term routine care.
Primary Care Physician Visit | At 14 months
  The number of participants that followed up with a primary care physician for a visit or to establish long-term routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Trapl, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Barbershops Local to Cleveland, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies results in publication.
Supporting Information: Study Protocol
Time Frame: Available immediately after publication with no end date.
Access Criteria: Researchers who provide a sound proposal.